CLINICAL TRIAL: NCT00926640
Title: A Phase I Study of Belinostat in Combination With Cisplatin and Etoposide in Adults With a Focus on Small Cell Lung Cancer and Other Cancers of Neuroendocrine Origin
Brief Title: A Phase I Study of Belinostat in Combination With Cisplatin and Etoposide in Adults With Small Cell Lung Carcinoma and Other Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090173; 09-C-0173
Record Dates: First submitted 2009-06-20; First posted 2009-06-23 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-04-20

CONDITIONS: Carcinoma Neuroendocrine; Small Cell Lung Carcinoma; Malignant Epithelial Neoplasms
Keywords: Solid Tumors; Histone deacetylase inhibitors; EP & Belinostat; Phase I; SCLC; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Small Cell Lung Carcinoma; Carcinoma | interventions — belinostat; Cisplatin; Etoposide

ARMS (3):
- 1 (Experimental): Belinostat dose escalation
  Interventions: Drug: Belinostat; Drug: Cisplatin; Drug: Etoposide
- 2 (Experimental): Belinostat UGT1A1 wild type/*28 variant
  Interventions: Drug: Belinostat; Drug: Cisplatin; Drug: Etoposide
- 3 (Experimental): Belinostat UGT1A1*60 or 2/3/4 variant
  Interventions: Drug: Belinostat; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Belinostat — 6 cycles of belinostat 400 mg/m2/24h X2 administered by CIV
Drug: Cisplatin — 6 cycles at 60mg/m2 IV on day 2
Drug: Etoposide — 6 cycles 80 mg/m2 IV daily X3 beginning day 2.

SUMMARY:
BACKGROUND:

* The histone deacetylase (HDAC) inhibitors are a novel class of anticancer agent. These agents lead to the increased acetylation of both histone and non-histone proteins, which leads to rapid cell death in many tumor models. It is thought that the cell death observed with this class of agents may be mediated, in part, through the selective acetylation of histone proteins resulting in increased expression of specific genes.
* For solid tumors in general, cell death in preclinical models has not translated to activity in patients. For this reason, studies increasingly have combined chemotherapy with HDAC inhibitors to achieve additive and potentially synergistic effects on cancer cells.
* This protocol will study a continuous infusion of the HDAC inhibitor belinostat in combination with cisplatin and etoposide for patients with advanced cancer.

OBJECTIVES:

* To determine a safe and tolerable phase 2 dose for the combination of belinostat with cisplatin and etoposide.
* Evaluate molecular markers of HDAC inhibition.

ELIGIBILITY:

* The protocol will be open to all patients with recurrent or advanced cancer (small-cell lung cancer and other advanced cancers) for whom standard therapy offers no curative potential.
* Age greater than or equal to 18 years
* ECOG Performance Status 0-2

DESIGN:

* The study will begin with belinostat 400 mg/m (2)/24h administered by continuous IV infusion on days 1 and 2, cisplatin at 80 mg/m (2) IV on day 2, and etoposide at 100 mg/m (2) IV daily times 3 on days 2 - 4. Dose escalation of belinostat will follow according to traditional 3 patient cohorts.
* Treatment schedule and dose escalation schemata.

DETAILED DESCRIPTION:
BACKGROUND:

* The histone deacetylase (HDAC) inhibitors are a novel class of anticancer agent. These agents lead to the increased acetylation of both histone and non-histone proteins, which leads to rapid cell death in many tumor models. It is thought that the cell death observed with this class of agents may be mediated, in part, through the selective acetylation of histone proteins resulting in increased expression of specific genes.
* For solid tumors in general, cell death in preclinical models has not translated to activity in patients. For this reason, studies increasingly have combined chemotherapy with HDAC inhibitors to achieve additive and potentially synergistic effects on cancer cells.
* This protocol will study a continuous infusion of the HDAC inhibitor belinostat in combination with cisplatin and etoposide for patients with advanced cancer.

OBJECTIVES:

* To determine a safe and tolerable phase 2 dose for the combination of belinostat with cisplatin and etoposide.
* Evaluate molecular markers of HDAC inhibition.
* To explore the results of administering the dose of belinostat based on the patients' UGT1A1 *28 or *60 genotype, which is a characteristic that may be associated with toxicity.

ELIGIBILITY:

* The protocol will be open to all patients with recurrent or advanced cancer (small-cell lung cancer and other advanced cancers) for whom standard therapy offers no curative potential.
* Age greater than or equal to 18 years
* ECOG Performance Status 0-2

DESIGN:

* The study will begin with belinostat 400 mg/m (2)/24h administered by continuous IV infusion on days 1 and 2, cisplatin at 60 mg/m(2) IV on day 2, and etoposide at 80 mg/ (2) IV daily times 3 on days 2 - 4. Dose escalation of belinostat will follow according to traditional 3 patient cohorts.
* With Amendment M, dosing will be based on UGT1A1 status, at either 400 mg/m(2) or

  600 mg/m(2)

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have histologic or cytologic confirmation of cancer for which there is no known standard therapy capable of extending life expectancy.
2. Patients must be greater than or equal to 4 weeks from cytotoxic chemotherapy, except greater than or equal to 6 weeks for mitomycin C or nitrosoureas, and greater than or equal to 8 weeks from prior UCN01; greater than or equal to 4 weeks from monoclonal antibody therapy (cetuximab, bevacizumab); greater than or equal to 4 weeks from prior experimental therapy; greater than or equal 2 weeks from radiation or hormonal therapy; greater than or equal to 2 weeks from sorafenib, sunitinib or temsirolimus treatment. Patients with prostate cancer may continue ongoing LhRH agonist therapy. Patients with bone metastases or hypercalcemia who began intravenous bisphosphonate treatment prior to study entry may continue this treatment while on study.
3. ECOG performance status 0-2.
4. Life expectancy of 3 months or greater.
5. Patients must have acceptable organ and marrow function as defined below:

   * absolute neutrophil count greater than or equal to 1,500/ mm(3)
   * platelets greater than or equal to 100,000/ mm(3)
   * total bilirubin less than or equal to 1.2 mg/dL (except patients with Gilbert's Syndrome)
   * AST (SGOT) and ALT(SGPT) less than or equal to 2.5 times institutional upper limit of normal
   * creatinine less than or equal to 1.5 times institutional upper limit of normal

   OR

   - creatinine clearance >50 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
6. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study, and for 3 months after study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
7. Age greater than or equal to 18 years.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Willing to comply with study procedures and follow-up.

EXCLUSION CRITERIA:

1. Patients who have not recovered (CTCAE less than or equal to grade 1) from adverse events due to prior treatments, except for alopecia or base stable grade 2 tinnitus (not interfering with ADL s) or stable grade 2 sensory neuropathy without pain or motor component, and not interfering with ADL s.
2. Patients may not have received more than 2 prior cytotoxic regimens.
3. Patients may not be receiving any other investigational agent with therapeutic anticancer intent.
4. Patients may not have taken another histone deacetylase inhibitor (i.e. valproic acid, vorinostat) for at least 2 weeks prior to enrollment.
5. Patients with history of CNS metastasis may not be enrolled on the study, unless control has been achieved with either radiation or surgical resection at least 3 months prior to enrollment on study.
6. Patients who have had radiation to the pelvis or other bone marrow-bearing sites will be considered on a case by case basis and may be excluded if the bone marrow reserve is not considered adequate (>25% of bone marrow).
7. Uncontrolled medical illness including, but not limited to ongoing or active infection, chronic or acute hepatitis, renal failure, symptomatic congestive heart failure, myocardial infarction unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. HIV-positive patients.
9. Patients with acute or chronic hepatitis.
10. Pregnant patients may not receive this experimental therapy.
11. Significant cardiovascular disease, myocardial infarction within the past 6 months, unstable angina, unstable arrhythmia or a need for anti-arrhythmic therapy (use of medication to control heart rate in patients with atrial fibrillation is allowed, if stable medication for at least last month prior to randomization and medication not listed as causing Torsade de Points), or evidence of acute ischemia on ECG.
12. Baseline prolongation of QT/QTc interval, i.e., defined as an average QTc interval > 450 msec; Long QT Syndrome; or the required use of concomitant medication that may cause Torsade de Pointes.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07-01; Primary Completion 2017-06-16 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Dose Limiiting Toxicity

SECONDARY OUTCOMES:
Markers of HDAC | End of treatment
Tumor response | Disease Progression
miRNA and CGH | End of treatment
Increased acetylation in PBMCs | End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Akerley W, McCoy J, Hesketh PJ, Goodwin JW, Bearden JD, Atkins JN, Chansky K, Crowley JJ, Gandara DR; SWOG. Gemcitabine and irinotecan for patients with untreated extensive stage small cell lung cancer: SWOG 0119. J Thorac Oncol. 2007 Jun;2(6):526-30. doi: 10.1097/JTO.0b013e318060d2dc. PMID 17545848
- [Background] Bevins RL, Zimmer SG. It's about time: scheduling alters effect of histone deacetylase inhibitors on camptothecin-treated cells. Cancer Res. 2005 Aug 1;65(15):6957-66. doi: 10.1158/0008-5472.CAN-05-0836. PMID 16061681
- [Background] Camphausen K, Scott T, Sproull M, Tofilon PJ. Enhancement of xenograft tumor radiosensitivity by the histone deacetylase inhibitor MS-275 and correlation with histone hyperacetylation. Clin Cancer Res. 2004 Sep 15;10(18 Pt 1):6066-71. doi: 10.1158/1078-0432.CCR-04-0537. PMID 15447991
- [Derived] Peer CJ, Hall OM, Sissung TM, Piekarz R, Balasubramaniam S, Bates SE, Figg WD. A population pharmacokinetic/toxicity model for the reduction of platelets during a 48-h continuous intravenous infusion of the histone deacetylase inhibitor belinostat. Cancer Chemother Pharmacol. 2018 Sep;82(3):565-570. doi: 10.1007/s00280-018-3631-7. Epub 2018 Jun 27. PMID 29951694